CLINICAL TRIAL: NCT02513823
Title: Effectiveness of Vitamin D Supplementation on Reducing Blood Pressure and Improving Endothelial Function of Pre-menopausal African American Women
Brief Title: Effectiveness of Vitamin D Supplementation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Reached power analysis goal and funds depleted
Sponsor: Texas Woman's University (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Carolyn Moore, Associate Professor, Texas Woman's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 11089
Record Dates: First submitted 2015-07-30; First posted 2015-08-03 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Elevated Blood Pressure; Endothelial Dysfunction
Keywords: blood pressure; vitamin D
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): 2,000 IU of vitamin D given to African American women for 10 weeks
  Interventions: Dietary Supplement: 2,000 International Units (IU)of vitamin D3

INTERVENTIONS:
Dietary Supplement: 2,000 International Units (IU)of vitamin D3 — 2,000 IU vitamin D taken daily for 10 weeks

SUMMARY:
This pilot study will examine the effectiveness of vitamin D supplementation on reducing blood pressure and improving endothelial function. Premenopausal African American women will be recruited. Participants will be instructed to record food intake for three days to estimate usual dietary intake at baseline and at the 10th week. At the baseline clinic visit a 10 week supply of vitamin D3 supplements (2,000 IU/day; Nature Made ®) will be given to participants and log sheets provided to record supplement intake. To answer the primary research questions, within subjects repeated measures analysis of variance (ANOVA) tests will be conducted to test if any differences in blood pressure, serum 25(OH)D concentrations, and RHI are statistically different after 10 weeks of supplementation with 2,000 IU/d of vitamin D. Exploratory multivariate linear regression models will be constructed to determine relationships between vitamin D status and vascular function parameters (blood pressure, RHI) before and after adjustment for age and BMI.

DETAILED DESCRIPTION:
This pilot study will examine the effectiveness of vitamin D supplementation on reducing blood pressure and improving endothelial function. If results of the pilot study are favorable, findings will be used to design a possibly larger study to confirm results. Premenopausal African American women (n = 40) will be recruited. All participant study visits will be held at the Houston Methodist Internal Medicine Clinic or at the TWU Nutrition Laboratory. African American women will be recruited who are not taking hypertensive medications, have average blood pressure measurements < 140/90 mmHg, are not pregnant or planning on becoming pregnant in the next three months, or who are not lactating.

Enrollment Visit The day prior to the enrollment visit potential subjects will fast overnight and refrain from consuming any caffeinated products, vitamins, or medications that may affect vascular tone and refrain from smoking. the investigators will explain the 10 week study design and obtain participant consent. Testing will be performed in the morning with start times between 8 and 10:00 a.m. In a quiet and temperature-controlled room (72° to 75° F), initial systolic and diastolic blood pressure measurements following 5 minutes of seated rest following the American Heart Association Blood Pressure Guidelines. The arm will be supported at heart level and neither participant nor observer will talk during the measurements. Three successive measurements will be collected with an automated oscillometric sphygmomanometer and the average of the last two measurements will be calculated. Any individual with an average blood pressure > 140/90 mmHg will be referred to their personal physician for follow up.

Consented participants with blood pressure readings <140/90 mmHg will be instructed to consume their usual diet for the next week and to complete a three-day diet record of two week days and one weekend. Instructions on how to record the dietary diary will be given. Food records will be used to estimate usual dietary intake for the baseline and 10 week time points. An appointment will be scheduled for the participant to return with completed food records to begin the intervention study. At the baseline clinic visit a 10 week supply of vitamin D3 supplements (2,000 IU/day; all the same lot; Nature Made ®) will be given to participants and log sheets provided to record supplement intake. In addition, participants will be instructed to avoid traveling to sunny locations for 10 weeks.

Baseline and 10 week clinic visits

Nutrient intake:

Three-day diet records will be collected during the baseline and 10 week clinic visits. Food records will be analyzed at TWU utilizing the University of Minnesota 2015 Nutrient Data System for Research. Total energy intake; percent calories from fat, protein and carbohydrates; and intake of vitamins A, C, D, E and beta carotene will be estimated from food records.

Blood pressure measurements:

Participants will fast overnight and refrain from consuming any caffeinated products, vitamins, medications that may affect vascular tone, or smoking. Testing will be performed in the morning with start times between 8 and 10:00 a.m. In a quiet and temperature-controlled room (72° to 75° F), initial systolic and diastolic blood pressure measurements will be taken following 5 minutes of seated rest following the American Heart Association Blood Pressure Guidelines. The arm will be supported at heart level and neither participant nor observer will talk during the measurements. Three successive measurements will be collected with an automated oscillometric sphygmomanometer and the average of the last two measurements will be calculated.

Body fat and adiposity measures:

Anthropometric and body fat distribution assessments will be performed. Height and weight will be measured. Percent body fat will be determined by bioelectric impedance (Tanita BF-350). Body mass index (BMI) will be calculated as weight in kilograms (kg) divided by height squared (m2).

Endothelial pulse amplitude measurements:

Pulse amplitude tonometry (PAT) will be measured with the EndoPAT 2000 (Itamar Medical Ltd) which records digital pulse wave amplitude (PWA) using fingertip plethysmography (16). The Endo-PAT finger probe consists of a thimble-shaped sensor cap that imparts a uniform pressure field and exhibits a clamp-like effect on the entire surface of the distal phalanx and measured pulsatile volume changes. PWA is measured continuously during three phases: a quiet baseline period, 5-minute forearm occlusion, and reactive hyperemia following cuff release. Occlusion of the brachial artery is performed on the non-dominant upper arm. The continuous monitoring of blood volume reaching the finger tips allows the hyperemic response to be quantified as a ratio, comparing PWA from pre to post occlusion. A reactive hyperemia index (RHI) measures nitric-oxide dependent changes in vascular tone. The recordings from the non-occluded arm serve as a control for changes in overall physiological state. The Endo-PAT RHI index is defined as the ratio of the average PWS during the 1 minute period beginning after exactly 90 second to reactive hyperemia compared with the average pulse amplitude during the 210 second pre-occlusion baseline period. Endothelial dysfunction is classified as a RHI < 1.67 with average normal endothelial RHI values ranging between 1.7 and 2.0.

Vitamin D measurements:

Blood will be drawn by Houston Methodist Hospital laboratory for measurement of serum 25(OH)D concentrations by chemiluminescence immunoassay( Abbott Architect). Vitamin D deficiency will be defined as serum 25(OH)D levels less than 20 ng/mL (50 nmol/L) and vitamin D insufficiency as 21 to 29 ng/mL (50 to 80 nmol/L).

Statistical analyses:

Descriptive statistics, including means and standard deviations for continuous variables and frequencies and percentages for categorical variables, will be calculated for study variables. Age, BMI, blood pressure, serum 25(OH)D concentration, and RHI will be treated as continuous variables. Prior to conducting primary analyses, exploratory and preliminary analyses will be conducted to test the statistical assumptions of planned analyses. Specifically, these assumptions include normality, homogeneity of variance, equivalent group size, and data that is missing by random. In the event that any of these assumptions have been violated, the data will either be transformed to meet the parametric assumptions of planned analyses or non-parametric equivalencies will be conducted as an alternative. In addition, correlation analyses, including Pearson's product moment correlations for normally distributed variables and Spearman's rho for non-normally distributed variables, will be conducted to examine the variables for potentially collinear relationships, which may impact primary analyses.

To answer the primary research questions, within subjects repeated measures analysis of variance (ANOVA) tests will be conducted to test if differences in blood pressure, serum 25(OH)D concentrations, and RHI are statistically different after 10 weeks of supplementation with 2,000 IU/d of vitamin D. Furthermore, exploratory multivariate linear regression models will be constructed to determine relationships between vitamin D status and vascular function parameters (blood pressure, RHI) before and after adjustment for age and BMI. All statistical analyses will be performed using Statistical analyses SPSS (version 19; SPSS IBM) and p < 0.05 will be used to determine statistical significance.

A priori power analyses was conducted using G*Power (v. 3.0.10) in order to determine an adequate sample size to detect statistical significance if significance in fact exists. In order to obtain a desired level of power at .80, estimating a moderate effect size (.25) and an alpha level of .05, a total of 22 participants will be needed to to ensure a statistically significant increase in serum 25(OH)D concentrations. Accounting for attrition of approximately 15%, a total of 25 participants will be recruited. Repeated measures-ANOVAs will be utilized to detect significant changes across the following outcome variables: serum 25(OH)D, blood pressure, and RHI. As such, a total of 25 participants should be sufficient to detect significance if significance in fact exists across all planned analyses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pre-menomausal African American women

Exclusion Criteria:

* History of elevated blood pressure >140/90 mm Hg
* Pregnant or planning to become pregnant in the next three months
* Lactating
* Known Crohn's
* Inflammatory bowel disease
* Previous bowel resections
* Bariatric surgeries, or psoriasis
* Artificial or long fingernails they do not want to cut for testing
* Regularly taking medications that might affect endothelial function such as anti-inflammatory medications, statins, anti-hypertensive medication, daily aspirin, non-SSRI psychotropic medication, and dietary supplements including vitamin D supplements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2016-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Moore, PHD, RD, LD, Principal Investigator — Methodist Hosptial
Locations (1):
- Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 27
Completed | 22
Not Completed | 5
Not completed — Lost to Follow-up | 4
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Vitamin D Supplementation on Reducing Blood Pressure
Description: Changes in systolic and diastolic blood pressure will be measured at baseline and following vitamin D supplementation for 10 weeks in African American healthy pre-menopausal women
Time Frame: Baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention
Number analyzed (Participants) | 22
mmHg
  SPB at Baseline | 124 (12)
  SBP at 10 Weeks | 125 (10)
  DBP at baseline | 79 (11)
  DBP at 10 weeks | 81 (10)

2. Secondary Outcome: Effectiveness of Vitamin d Supplementation on Improving Endothelial Function
Description: Changes of endothelial function at baseline and following 10 weeks of vitamin D supplementation as measured by pulse amplitude tonometry (PAT) fingertip plethysmography. Endothelial dysfunction was classified as a Reactive Hyperemic Index (RHI) of < 1.67 . RHI scale typical ranges from 1.0 to 3.0.
Time Frame: Baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 22
units on a scale
  Reactive Hyperemia Index Baseline | 2.1 (0.6)
  Reactive Hyperemia Index 10 Weeks | 2.0 (0.5)

ADVERSE EVENTS:
Time Frame: 10 weeks over the vitamin D supplementation period
Description: Participants could contact the investigators with questions or concerns.
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No